CLINICAL TRIAL: NCT03875976
Title: Randomised Controlled Study Comparing Fast Track and Standard Care Protocol on Functional Outcomes and Hospital Stay Of Total Hip Arthroplasty
Brief Title: Total Hip Arthroplasty: Fast Track Protocol is the Future?
Acronym: FastTrack-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Dante Dallari, MD, MD, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11269
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Hip Osteoarthritis; Arthropathy of Hip
Keywords: fast track care; total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: The study aims to evaluate the effectiveness of a fast track protocol , which consists of an innovative analgesic therapy scheme and a rapid rehabilitation protocol, and a standard care protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Track Protocol (Active Comparator): Patients treated using Fast Track Care Protocol
  Interventions: Procedure: Fast Track Protocol
- Standard Protocol (Active Comparator): Patients treated using Standard Care Protocol
  Interventions: Procedure: Standard Care Protocol

INTERVENTIONS:
Procedure: Fast Track Protocol — Fast Track Care consists in educational preoperative preparation for patients, particular strategies for controlling pain and intensive early rehabilitation protocol
  Arms: Fast Track Protocol
Procedure: Standard Care Protocol — Standard Care Protocol consists in the same surgical intervention without educational preoperative preparation for patients and intensive early rehabilitation protocol
  Arms: Standard Protocol

SUMMARY:
Fast-track total hip arthroplasty (THA) is a well-established concept including optimized logistics and evidence-based treatment, focusing on minimizing surgical stress and improved post-operative recovery. The aim of this protocol is to compare the standard care and fast track total hip arthroplasties in terms of functional and subjective outcomes, hospital staying, number of transfusions and analgesic consumption.

DETAILED DESCRIPTION:
The aim of this protocol is to compare standard care and fast track total hip arthroplasties. The fast track care consists of:

* preoperative educational lesson in which orthopedic surgeon, anesthesiologist and physiotherapist illustrate the operative and post operative path to the patients
* antalgic protocol administered only orally
* early rehabilitation care. The day of the surgical operation, the physiotherapist helps the patient reach the upright position. The standard care consists of usual antalgic and physiotherapy post-operative care:
* Antalgic protocol consist in intravenous drugs
* the first physiotherapy session is the day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by hip osteoarthritis, eligible for primary total hip arthroplasty
* BMI < 32
* Time up ang go test </= 12 seconds
* American Society of Anesthesiologists physical status classification system (ASA) </= 2
* preoperative hemoglobin (HB) >13 g/dl
* patients eligible for spinal anesthesia
* presence of a care-giver

Exclusion Criteria:

* psychiatric diseases
* preoperative use of crutches
* ASA > 3
* preoperative HB < 13 g/dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Early functional outcomes | Third post operative day
  Early functional outcomes are collecting using Lowa Level of Assistance(ILOA) during the third post-operative day.
  This scale is able to provide data on the autonomy reached by the patient in the first postoperative period going to investigate five main motor activities (get up from supine to seated, from sitting to standing position, walk around, take three steps, the speed of walking). The total score can vary from 0 to 56, where 56 indicates worst functional results.

SECONDARY OUTCOMES:
hospital staying | Third post operative day
  The collection of hospital stay for each patient. The fast track expecting hospital stay is three days.
Incidence of early major complications | Third day after surgery
  The collection of acute infection and early fracture
Number of transfusions | Third day after surgery
  the collection of number of transfusions during hospital staying
Analgesic consumption | Third day after surgery
  The request for analgesic rescue in relation to fast track standard analgesic scheme
Harris Hip Score (HHS) at 6 weeks | 6 weeks after surgery
  The collection of functional outcomes HHS at 6 weeks. The HHS is made of four subscales. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points). The higher scores representing less dysfunction and better outcomes.
Harris Hip Score (HHS) at third month | third month after surgery
  The collection of functional outcomes HHS at third month. The HHS is made of four subscales. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points). The higher scores representing less dysfunction and better outcomes
Harris Hip Score (HHS) at sixth month | sixth month after surgery
  The collection of functional outcomes HHS at sixth month. The HHS is made of four subscales. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points). The higher scores representing less dysfunction and better outcomes
Harris Hip Score (HHS) at twelfth month twelfth | twelfth month after surgery
  The collection of functional outcomes HHS at twelfth month. The HHS is made of four subscales. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points). The higher scores representing less dysfunction and better outcomes
WOMAC at 6 weeks | 6 weeks after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher scores representing less outcomes.
WOMAC at third month | Third month after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher scores representing less outcomes.
WOMAC at sixth month | Sixth month after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher scores representing less outcomes.
WOMAC at twelfth month | twelfth month after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher scores representing less outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dante Dallari, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Derived] Rocchi M, Stagni C, Govoni M, Mazzotta A, Vivarelli L, Orlandi Magli A, Perrone M, Benedetti MG, Dallari D. Comparison of a fast track protocol and standard care after hip arthroplasty in the reduction of the length of stay and the early weight-bearing resumption: study protocol for a randomized controlled trial. Trials. 2021 May 17;22(1):348. doi: 10.1186/s13063-021-05314-5. PMID 34001185